CLINICAL TRIAL: NCT03256032
Title: Prevalence and Factors Associated With Postoperative Hypothermia Among Patients Undergoing Anaesthesia and Surgery in Mulago National Referral Hospital
Brief Title: Prevalence and Factors Associated With Postoperative Hypothermia in Mulago Hospital
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: POSTOP HYPOTHERMIA MULAGO
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Post Operative Hypothermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Patient's sublingual temperature was measured postoperatively on entry to the recovery room.

DETAILED DESCRIPTION:
Adult patients who underwent non-neurological and non-cardiac surgery had their sublingual temperature measured postoperatively on entry to the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* All patients of 18 years and above, undergoing surgery and anaesthesia lasting longer than 30minutes.
* All patients of 18 years and above, undergoing elective and emergency non cardiac and non-neurological operations in Mulago National Referral Hospital.

Exclusion Criteria:

* Patients with contraindications to measurement of sublingual temperature

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery and anaesthesia at Mulago National Referral Hospital who meet the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative hypothermia | July 2016 to February 2017
  Sublingual temperature at entry to the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Emoru, Principal Investigator — MakCHS

IPD SHARING:
Plan to Share IPD: Undecided